CLINICAL TRIAL: NCT04112589
Title: A Multicenter, Prospective, Non-randomized, Phase I-II Trial to Assess the Efficacy and Safety of the Combination of Oral Quizartinib and the FLAG-IDA Chemotherapy Regimen in First Relapsed/Refractory Acute Myeloid Leukemia (R/R AML) Patients
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of the Combination of a Drug Call Quizartinib With Chemotherapy (FLAG-IDA) in Patients With Acute Myeloid Leukemia That Has Not Responded to the First Treatment or That Has Returned After the First Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry); Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FLAG-QUIDA
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib; fludarabine; Cytarabine; Idarubicin

STUDY DESIGN:
Intervention Model Description: The study consists of a dose escalation-dose finding part (phase I) and a phase II part.
  Subjects will have an induction of 1 cycle, by an alloSCT (allogeneic hematopoietic stem cell transplantation) in CR/CRi, when possible, with up to 3 optional HiDAC (high dose Cytarabine ) consolidation cycles. All patients in CR/CRi will receive a maintenance schedule (12 months, 12 cycles).
  The phase I portion will progress from starting level dose 1 (40mg 14 days) to level dose 2 (60 mg 14 days). De-escalation to level dose -1 (60mg 7 days) or level dose -2 (40mg 7 days) may be necessary to be explored.
  Once the RP2D is established, the phase II will start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Level dose 1 - 40mg, 14 days (Experimental): Patients will receive an induction cycle (40mg Quizartinib for 14 days) followed by 1-3 consolidation cycles (Quizartinib at day 6) [with or without allogenic stem cell transplantation]- Responders will have 12 months maintenance starting at 30mg/day Quizartinib will be increased to 60 mg/day after 15 days if appropriate.
  Interventions: Drug: Quizartinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: glycosylated G-CSF
- Level dose 2 - 60mg, 14 days (Experimental): Patients will receive an induction cycle (60mg Quizartinib for 14 days) followed by 1-3 consolidation cycles (Quizartinib at day 6) [with or without allogenic stem cell transplantation]- Responders will have 12 months maintenance starting at 30mg/day Quizartinib will be increased to 60 mg/day after 15 days if appropriate.
  Interventions: Drug: Quizartinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: glycosylated G-CSF
- Level dose -1 - 60mg 7days (Experimental): Patients will receive an induction cycle (60mg Quizartinib for 7 days) followed by 1-3 consolidation cycles (Quizartinib at day 6) [with or without allogenic stem cell transplantation]- Responders will have 12 months maintenance starting at 30mg/day Quizartinib will be increased to 60 mg/day after 15 days if appropriate.
  Interventions: Drug: Quizartinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: glycosylated G-CSF
- Level dose -2 - 40mg 7 days (Experimental): Patients will receive an induction cycle (40mg Quizartinib for 7days) followed by 1-3 consolidation cycles (Quizartinib at day 6) [with or without allogenic stem cell transplantation]- Responders will have 12 months maintenance starting at 30mg/day Quizartinib will be increased to 60 mg/day after 15 days if appropriate.
  Interventions: Drug: Quizartinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Idarubicin; Drug: glycosylated G-CSF

INTERVENTIONS:
Drug: Quizartinib — Quizartinib at different doses in the phase I (40mg-14 days; 60mg-14 days; 60mg-7days, 40mg-7days). RP2D in the phase II part.
Drug: Fludarabine — 30 mg/m2 intravenous days 1 to 4 of the cycle
Drug: Cytarabine — 2 g/m 2 intravenous days 1 to 4 (1 g/m2 in patients older than 59) of the cycle
Drug: Idarubicin — 10 mg/ 2 intravenous days 1 to 3 of the cycle
Drug: glycosylated G-CSF — daily dose of 300 mcg/m 2 , from day -1 until day 5 of the cycle

SUMMARY:
This is a multicenter, prospective, non-randomized, Phase I-II trial to assess the efficacy and safety of the combination of oral quizartinib and FLAG-IDA chemotherapy schedule (FLAG-QUIDA regimen) in first relapsed/refractory AML (acute myeloid leukemia) patients.

DETAILED DESCRIPTION:
Patients of approximately 20 sites (in Spain and Portugal) will receive FLAG-QUIDA regimen followed by transplantation, when possible, with up to 3 optional consolidation cycles. All patients in CR/CRi (complete remission / complete remission with incomplete hematologic recovery) will receive a maintenance schedule.

A Phase I (dose escalation) will be performed at 40 mg x 14 days of quizartinib in the first 3 patients, and if no dose-limiting toxicity (DLT) is observed, the next cohort of patients will receive 60 mg x 14 days. There is also the possibility of de-escalation cohorts at 60 mg x 7 days and at 40 mg x 7 days. Patients participating in the Phase I will receive the allocated dose level, and therefore, they must not receive strong CYP3A4 inhibitors concomitantly with quizartinib The Phase II will include 68 patients treated at the RP2D (recommended phase 2 dose). A 1-year maintenance schedule starting at 30 mg will be increased to 60 mg/day if appropriate.

Patients will be followed up for a minimum period of 1 year since the first visit of the last patient included.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with national, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure. Informed consent form must be signed by the patient and the Investigator.
2. Patients aged ≥ 18 years old and ≤70 years old at the time of screening.
3. First R/R AML defined as:

   * First relapse after frontline intensive chemotherapy (with or without prior alloSCT), irrespectively of the duration of the first CR. Patients previously treated with a FLT3 inhibitor different from quizartinib, can be included.
   * First refractory disease (defined as patients not achieving at least a PR after first induction cycle and/or not achieving CR/CRi after first 2 cycles). Patients previously treated with a FLT3 inhibitor different from quizartinib, can be included.
4. Non-APL AML.
5. Considered for intensive approach as per Investigator judgment.
6. ECOG 0-2.
7. No contraindications for quizartinib.
8. No contraindications for intensive chemotherapy.
9. No severe organ function abnormalities.
10. No active relevant GVHD.
11. For the Phase II, FLT3-ITD patients will represent 50% of the study cohort (FLT3-TKD are not excluded but included in the FLT3-ITD-WT group).
12. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use reliable methods of contraception upon enrollment, during the treatment period and for 6 months following the last dose of investigational drug or cytarabine, whichever is later.
13. Male patients must use a reliable method of contraception (if sexually active with a female of child-bearing potential) upon enrollment, during the treatment period, and for 6 months following the last dose of investigational drug or cytarabine, whichever is later.

Exclusion Criteria:

1. Patients with genetic diagnosis of acute promyelocytic leukemia.
2. Blastic phase of bcr/abl chronic myeloid leukemia.
3. Patients with other neoplastic disease, for whom the Investigator has clinical suspicion of active disease at the time of enrollment. Note: Patients with adequately treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia are eligible for this study. Hormonal or adjuvant therapies will be allowed for breast cancer or prostate cancer if they are on a stable dose for at least 2 weeks prior to first dose.
4. Presence of any severe psychiatric disease or physical condition/comorbidity that, according to the physician´s criteria, contraindicates the inclusion of the patient in the clinical trial
5. Serum creatinine ≥ 250 μmol/l (≥ 2.5 mg/dL) (unless it is attributable to AML activity).
6. Bilirubin, alkaline phosphatase, or SGOT >3 times the upper normal limit (unless it is attributable to AML activity).
7. Uncontrolled or significant cardiovascular disease, including any of the following:

   * Symptomatic bradycardia of less than 50 beats per minute, unless the subject has a pacemaker.
   * QTcF >450 ms at screening. Note: QTcF will be derived from the mean of triplicate readings.
   * Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome)
   * History of clinically relevant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes).
   * History of second- (Mobitz II) or third-degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker).
   * History of uncontrolled angina pectoris or myocardial infarction within 6months prior to Screening.
   * History of New York Heart Association Class 3 or 4 heart failure.
   * Complete left bundle branch block.
   * Right bundle branch and left anterior hemiblock (bifascicular block)
   * Infarction (MI) within 3 months.
   * Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥ 110 mmHg
   * A previously known left ventricle ejection fraction <45%
8. Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; however, prophylactic use of these agents is acceptable even if parenteral.
9. Active hepatitis B or hepatitis C infection.
10. Previously known and documented human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this study).
11. Active acute or chronic GVHD requiring prednisone >10 mg or equivalent corticosteroid daily
12. Any patients with known significant impairment in gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of quizartinib
13. History of hypersensitivity to any excipients in the quizartinib tablets.
14. Females who are pregnant or breastfeeding.
15. Isolated extramedullary R/R AML.
16. Only applicable to patients screened after the first cohort of 34 patients of the Phase II has been achieved (e.g., FLT3-ITD negative): patients must have a confirmation of FLT3-ITD status at relapse, and this must correspond to the non-achieved cohort (e.g. FLT3-ITD positive).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
RP2D finding | 1 cycle (4 weeks)
  Maximum Tolerated dose of the combination of quizartinib a FLAG-IDA regimen
Rate CR/CRi | 3 years
  To assess the rate of CR/CRi after one cycle of FLAG-QUIDA

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  time from the first documentation of remission to the documentation of disease recurrence or death
Overall survival (OS) | 3 years
  Number of days from randomization until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, MD, Study Director — Trial Coordinator, Institution Contact
Locations (20):
- Spain (20):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Institut Català D'Oncologia-Hospital Germans Trias I Pujol, Badalona
  - Institut Català D'Oncologia-Hospital Duran I Reynals, Bellvitge
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - ICO Girona - Hospital Josep Trueta, Girona
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera
  - Complejo Hospitalario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Universitario Virgen Del Rocío, Seville
  - Hospital Universitari Joan Xxiii de Tarragona, Tarragona
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Forman SJ, Rowe JM. The myth of the second remission of acute leukemia in the adult. Blood. 2013 Feb 14;121(7):1077-82. doi: 10.1182/blood-2012-08-234492. Epub 2012 Dec 14. PMID 23243288
- [Background] Estey EH. Treatment of relapsed and refractory acute myelogenous leukemia. Leukemia. 2000 Mar;14(3):476-9. doi: 10.1038/sj.leu.2401568. PMID 10720145
- [Background] Yavuz S, Paydas S, Disel U, Sahin B. IDA-FLAG regimen for the therapy of primary refractory and relapse acute leukemia: a single-center experience. Am J Ther. 2006 Sep-Oct;13(5):389-93. doi: 10.1097/01.mjt.0000181690.21601.09. PMID 16988532
- [Background] Pastore D, Specchia G, Carluccio P, Liso A, Mestice A, Rizzi R, Greco G, Buquicchio C, Liso V. FLAG-IDA in the treatment of refractory/relapsed acute myeloid leukemia: single-center experience. Ann Hematol. 2003 Apr;82(4):231-5. doi: 10.1007/s00277-003-0624-2. Epub 2003 Mar 15. PMID 12707726
- [Background] de la Rubia J, Regadera A, Martin G, Cervera J, Sanz G, Martinez J, Jarque I, Garcia I, Andreu R, Moscardo F, Jimenez C, Molla S, Benlloch L, Sanz M. FLAG-IDA regimen (fludarabine, cytarabine, idarubicin and G-CSF) in the treatment of patients with high-risk myeloid malignancies. Leuk Res. 2002 Aug;26(8):725-30. doi: 10.1016/s0145-2126(02)00003-6. PMID 12191567
- [Background] Kim H, Park JH, Lee JH, Lee JH, Joo YD, Lee WS, Bae SH, Mo Ryoo H, Lee KH; Cooperative Study Group A for Hematology. Continuous infusion of intermediate-dose cytarabine and fludarabine with idarubicin for patients younger than 60 years with resistant acute myeloid leukemia: a prospective, multicenter phase II study. Am J Hematol. 2009 Mar;84(3):161-6. doi: 10.1002/ajh.21351. PMID 19195034
- [Background] Bergua JM, Montesinos P, Martinez-Cuadron D, Fernandez-Abellan P, Serrano J, Sayas MJ, Prieto-Fernandez J, Garcia R, Garcia-Huerta AJ, Barrios M, Benavente C, Perez-Encinas M, Simiele A, Rodriguez-Macias G, Herrera-Puente P, Rodriguez-Veiga R, Martinez-Sanchez MP, Amador-Barciela ML, Riaza-Grau R, Sanz MA; PETHEMA group. A prognostic model for survival after salvage treatment with FLAG-Ida +/- gemtuzumab-ozogamicine in adult patients with refractory/relapsed acute myeloid leukaemia. Br J Haematol. 2016 Sep;174(5):700-10. doi: 10.1111/bjh.14107. Epub 2016 Apr 26. PMID 27118319
- [Background] Cortes J, Perl AE, Dohner H, Kantarjian H, Martinelli G, Kovacsovics T, Rousselot P, Steffen B, Dombret H, Estey E, Strickland S, Altman JK, Baldus CD, Burnett A, Kramer A, Russell N, Shah NP, Smith CC, Wang ES, Ifrah N, Gammon G, Trone D, Lazzaretto D, Levis M. Quizartinib, an FLT3 inhibitor, as monotherapy in patients with relapsed or refractory acute myeloid leukaemia: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2018 Jul;19(7):889-903. doi: 10.1016/S1470-2045(18)30240-7. Epub 2018 May 31. PMID 29859851
- [Background] Cortes JE, Kantarjian H, Foran JM, Ghirdaladze D, Zodelava M, Borthakur G, Gammon G, Trone D, Armstrong RC, James J, Levis M. Phase I study of quizartinib administered daily to patients with relapsed or refractory acute myeloid leukemia irrespective of FMS-like tyrosine kinase 3-internal tandem duplication status. J Clin Oncol. 2013 Oct 10;31(29):3681-7. doi: 10.1200/JCO.2013.48.8783. Epub 2013 Sep 3. PMID 24002496
- [Background] Cortes JE, Tallman MS, Schiller GJ, Trone D, Gammon G, Goldberg SL, Perl AE, Marie JP, Martinelli G, Kantarjian HM, Levis MJ. Phase 2b study of 2 dosing regimens of quizartinib monotherapy in FLT3-ITD-mutated, relapsed or refractory AML. Blood. 2018 Aug 9;132(6):598-607. doi: 10.1182/blood-2018-01-821629. Epub 2018 Jun 6. PMID 29875101
- [Background] Chen Y, Pan Y, Guo Y, Zhao W, Ho WT, Wang J, Xu M, Yang FC, Zhao ZJ. Tyrosine kinase inhibitors targeting FLT3 in the treatment of acute myeloid leukemia. Stem Cell Investig. 2017 Jun 2;4:48. doi: 10.21037/sci.2017.05.04. eCollection 2017. PMID 28607922
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Creutzig U, Kaspers GJ. Revised recommendations of the International Working Group for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in acute myeloid leukemia. J Clin Oncol. 2004 Aug 15;22(16):3432-3. doi: 10.1200/JCO.2004.99.116. No abstract available. PMID 15310791
- [Background] Montesinos P, Lorenzo I, Martin G, Sanz J, Perez-Sirvent ML, Martinez D, Orti G, Algarra L, Martinez J, Moscardo F, de la Rubia J, Jarque I, Sanz G, Sanz MA. Tumor lysis syndrome in patients with acute myeloid leukemia: identification of risk factors and development of a predictive model. Haematologica. 2008 Jan;93(1):67-74. doi: 10.3324/haematol.11575. PMID 18166787